CLINICAL TRIAL: NCT03779373
Title: Manual Versus Assisted Fluid Management in Patients Undergoing Major Abdominal and Orthopedic Surgery: A Randomized Controlled Trial
Brief Title: Assisted Fluid Management in Patients Undergoing Major Abdominal and Orthopedic Surgery
Acronym: AFM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of hospital when the study will be done. We will redo the clinical trial to have the good sponsor for the study.
Sponsor: Erasme University Hospital (Other)
Collaborators: APHP (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, Principal Investigator, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-A03365-50
Record Dates: First submitted 2018-12-16; First posted 2018-12-19 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Goal Directed Fluid Therapy

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EV1000 monitoring (Active Comparator): This group of patients will receive fluid administration during surgery based on a manual GDFT protocol actually in place in the department using the EV1000 monitoring device (Edwards Lifesciences, Irvine, USA)
  Interventions: Other: Use of a decision support system on the EV1000 monitor (AFM mode)
- EV1000 monioring with the decision (AFM) (Experimental): This group of patients will receive fluid administration during surgery based on a novel clinical decision support system for GDFT guidance using the EV1000 monitoring device (Edwards Lifesciences, Irvine, USA)
  Interventions: Other: Use of a decision support system on the EV1000 monitor (AFM mode)

INTERVENTIONS:
Other: Use of a decision support system on the EV1000 monitor (AFM mode) — The way to administer fluid is based on the same monitoring device but will differ by the way fluid is given ( following a manual GDFT protocol versus following recommendation from an active clinical deicsion support system for fluid administration called AFM (assisted fluid management)

SUMMARY:
This study will compare a group of patients managed with a manual GDFT protocol (using the EV1000 monitoring device; Edwards Lifesciences, Irvine, USA) to a group of patients managed using a decision support system for GDFT guidance (implemented on the same EV1000 monitoring) in patients undergoing major abdominal and orthopedic surgery.

DETAILED DESCRIPTION:
Many trials have indicated that goal-directed fluid therapy (GDFT) strategies may benefit high-risk surgical patients but these strategies are infrequently implemented. It has also been shown that without any goal or protocol for fluid resuscitation, large inter- and intra-provider variability exist and have been correlated with marked variations in patient outcomes. Even under ideal study conditions, strict adherence to GDFT protocols is hampered by the workload and concentration required for consistent implementation.Haemodynamic monitors and protocols alone do not enable optimal fluid titration to be provided consistently to all patients - there must also be appropriate and timely interpretation and intervention.

To address this problem of consistency and protocol adherence, a clinical decision support system, "Assisted Fluid Management" (AFM), has been designed to help ease some of the workload associated with GDFT protocol implementation. The AFM system (released on the European market in March 2017) may help increase GDFT protocol adherence while leaving direction and guidance in the hands of the care providers. This system can suggest fluid bolus administration, analyse the effects of the bolus, and continually re-assess the patient for further fluid requirements.

A recent published study demonstrated that the implementation of the AFM for GDFT guidance resulted in a significantly longer period during surgery with a SVV <13% with a reduced total amount of fluid administered without any difference in postoperative complications. Therefore the goal of this randomized controlled trial is to compare a manual GDFT approach ( standard of care actually in the department) versus an Assisted fluid management approach (using the AFM mode) on the incidence of minor postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients in the operating room scheduled for a major abdominal & orthopedic surgery requiring a cardiac output monitoring (EV1000).
* Written informed consent received before surgery.

Exclusion Criteria:

* Minor Patients.
* No french speaking.
* Atrial fibrillation or severe arythmia.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
composite criteria of minor postoperative complications | 30 days postsurgery
  This composite score includes 8 items :
  1. postoperative nausea and vomiting
  2. delirium and confusion
  3. Infection of surgical site
  4. urinary infection
  5. acute kidney injury (KDIGO I & II classiciation)
  6. paralytic ileus
  7. other infection (skin, catheter, unknown etc)
  8. Readmission to the hospital within 30 days postoperative

SECONDARY OUTCOMES:
Percentage of Time spent during the procedure with a stroke volume variation < 13% | Postoperative day 1
  Percentage of Time spent during the procedure with a stroke volume variation < 13%
Percentage of Time spent during the procedure with a Cardiac index >2.5l/min/m2 | Postoperative day 1
  Percentage of Time spent during the procedure with a Cardiac index >2.5l/min/m2
composite criteria of major postoperative complications | 30 days postsurgery
  This composite score includes 14 items :
  1. stoma dehiscence
  2. Peritonitis
  3. Sepsis
  4. wound dehiscence
  5. bleeding requiring a redo surgery
  6. pulmonary embolism
  7. pulmonary edema
  8. Pneumonia
  9. acute coronary syndrome
  10. atrial fibrillation
  11. stroke
  12. Dialysis
  13. non scheduled redo surgery
  14. 30days mortality (all causes)
cardiac index over the procedure | Postoperative day 1
  average cardiac index over the surgery
stroke volume over the procedure | Postoperative day 1
  average stroke volume over the procedure
stroke volume variation over the procedure | Postoperative day 1
  average stroke volume variation over the procedure
Total Fluid received during the procedure | Postoperative day 1
  amount of fluid received during surgery
Net fluid balance | Postoperative day 1
  Net fluid balance at the end of the ICU stay
Postoperative acute care unit or intensive care unit length of stay | 30 days postsurgery
  Postoperative acute care unit or intensive care unit length of stay
Hospital length of stay | 30 days postsurgery
  hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Duranteau, PhD, Study Director — Bicetre Hospital; APHP BICETRE, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Joosten Alexandre, Paris, Kremlin Bicetre, France

IPD SHARING:
Plan to Share IPD: No